CLINICAL TRIAL: NCT02368860
Title: Phase I Trial of OXIRI [Oxaliplatin (O), Xeloda (X) and Irinotecan (I)] Treatment in Patients With Advanced and/or Metastatic Pancreatic Adenocarcinoma
Brief Title: OXIRI [Oxaliplatin (O), Xeloda (X) and Irinotecan (I)] in Pancreatic Adenocarcinoma
Acronym: OXIRI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-13-01
Record Dates: First submitted 2015-01-29; First posted 2015-02-23 (Estimated); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Irinotecan; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OXIRI (Experimental): OXIRI regimen: oxaliplatin, irinotecan, capecitabine
  Interventions: Drug: oxaliplatin, irinotecan, capecitabine

INTERVENTIONS:
Drug: oxaliplatin, irinotecan, capecitabine — fixed doses of intravenous oxaliplatin 50 mg/m2, and intravenous irinotecan administered on days 1 and 8 in a 21 day-cycle while xeloda will be administered daily at around midnight from day 1 to day 14
  Other Names: Eloxatin, Camptosar, CPT-11, Xeloda

SUMMARY:
This is an exploratory Phase I study is to assess the safety and tolerability of the OXIRI regimen [oxaliplatin (O), xeloda (X) and irinotecan (I)] and to evaluate for preliminary evidence of efficacy, in patients with advanced and/or metastatic pancreatic adenocarcinoma. The investigators hypothesize that 2 of 3 weekly doses of oxaliplatin and genotype directed-dosing of irinotecan in combination with chronomodulated capecitabine (xeloda) administered continuously will be more tolerable than the FOLFIRINOX regimen (folinic acid, fluorouracil, irinotecan and oxaliplatin) while maintaining anti-tumour activity.

DETAILED DESCRIPTION:
This study comprises a dose escalation phase using 3+3 design to determine the safety, tolerability and pharmacokinetics of the OXIRI regimen and an expansion phase to further evaluate the MTD and to determine early signs of efficacy.

Eligible patients will receive a novel chemotherapeutic regimen (OXIRI regimen) with xeloda being administered in a chronomodulated fashion and the dose of irinotecan being guided by the UGT1A1*28 and UGT1A1*6 genotype status of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 21 to 75 years of age
2. A histopathologically or cytological confirmed diagnosis of locally advanced and/or metastatic PDAC that is unresectable
3. Measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) ver 1.1 criteria
4. Life expectancy of at least 12 weeks
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
6. Adequate hematologic function (neutrophils count ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L)
7. Adequate hepatic function (total bilirubin ≤ 1.5 x the upper limits of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN
8. Adequate renal function (calculated creatinine clearance > 50 mL/min)
9. Able to give informed consent
10. Toxicity related to previous radiotherapy or chemotherapy resolved to ≤ Grade 1

Exclusion Criteria:

1. History of prior malignancy except non-melanoma skin cancer within the last 5yrs
2. Uncontrolled central nervous system (CNS) metastases or carcinomatous meningitis
3. Uncontrolled concomitant medical illnesses (e.g. hypertension, myocardial infarct, heart failure, ventricular arrhythmia, diabetes, severe infection)
4. Major surgery within four weeks prior to study treatment
5. Patients on chronic immunosuppressive therapy
6. Pregnant or breast-feeding female patients
7. On anticoagulant therapy with vitamin K antagonists.
8. Dose-escalation cohort:

   * Patients homozygous for uridine diphosphate glucuronosyltransferase (UGT)1A1*6/*6 or UGT1A1*28/*28
   * Previous oxaliplatin or irinotecan chemotherapy
   * Treatment with any of the following anti-cancer therapies prior to the first dose of OXIRI within the stated timeframes

     * Cyclical chemotherapy within a period of time that is shorter than the cycle length used for that treatment. Exception for weekly chemotherapy regimens, where a minimum of 2 week washout from the last dose is required.
     * Biological therapy (e.g., antibodies) within a period of time that is ≤ 5 t1/2 or ≤ 4 weeks, whichever is shorter, prior to starting study drug
     * Continuous or intermittent small molecule therapeutics within a period of time that is ≤ 5 t1/2 or ≤ 4 weeks (whichever is shorter) prior to starting study drug
     * Any other investigational agents within a period of time that is ≤ 5 t1/2 or less than the cycle length used for that treatment or ≤ 4 weeks (whichever is shortest) prior to starting study drug
     * Wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug
9. Dose-expansion cohort:

   * Previous chemotherapy or radiotherapy

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-09-17 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of the OXIRI regimen as measured by the frequency of significant adverse events incurred by the participants, using CTCAE ver. 4 grading system | from first dose to 30 days after last dose
  The safety and tolerability of the regimen will be assessed when the patient is on treatment and till 30 days after treatment.

SECONDARY OUTCOMES:
Maximum tolerated dose (MTD) of capecitabine when administered in a continuous chronomodulated fashion with genotype-directed dosing of irinotecan and metronomic dosing of oxaliplatin, using a conventional 3+3 design | 2 years
Recommended Phase II dose (RP2D) of the OXIRI regimen which is the MTD | 2 years
Pharmacokinetics analysis of capecitabine | cycle 1 day 1
  Plasma level of capecitabine, its intermediary metabolites (5'-deoxy-5-fluorocytidine [DFCR] and 5'- deoxy-5- fluorouridine [DFUR]) and 5FU will be measured at multiple time points on C1D1
Pharmacokinetics analysis of Irinotecan | cycle 1 day 1
  Plasma level of Irinotecan, SN-38 (active metabolite of irinotecan) and SN-38G will be measured at multiple time points on C1D1
Efficacy of OXIRI as measured by response evaluation criteria in solid tumours (RECIST) version 1.1 | 3 years

OTHER OUTCOMES:
Circulating tumour cells (CTCs) analysis | at pre-treatment, Day 1 of each cycle and during response evaluation by imaging
  CTC characterization, and the changes of CTCs number and their relationship to changes in serum CA19-9 levels, tumour response on imaging etc. will be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew CH Ng, Dr, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore